CLINICAL TRIAL: NCT04889495
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multicenter, Post-marketing Surveillance to Assess the Safety and Effectiveness of Zirabev in Domestic Patients With Non-small Cell Lung Cancer, Metastatic Colorectal Cancer, Metastatic Breast Cancer, Advanced or Metastatic Kidney Cancer, Cervical Cancer, Epithelial Ovarian Cancer, Fallopian Tube Cancer, Primary Peritoneal Cancer or Glioblastoma Multiforme.
Brief Title: A Post-marketing Surveillance to Assess the Safety and Effectiveness of Zirabev in Domestic Patients With Various Cancer
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn due to global supply chain issue. Zirabev was not launching in Korea.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7391012; NCT04889495 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer; Metastatic Colorectal Cancer; Metastatic Breast Cancer; Metastatic Kidney Cancer; Cervical Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Zirabev
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms; Kidney Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants receiving Zirabev: Participants receiving Zirabev
  Interventions: Drug: Zirabev

INTERVENTIONS:
Drug: Zirabev — Bevacizumab biosimilar

SUMMARY:
This is a prospective, single-arm, open-label, non-interventional, multicenter, post-marketing surveillance to assess the safety and effectiveness of Zirabev(Bevacizumab biosimilar) in domestic patients with non-small cell lung cancer, metastatic colorectal cancer, metastatic breast cancer, advanced or metastatic kidney cancer, cervical cancer, epithelial ovarian cancer, fallopian tube cancer, primary peritoneal cancer or glioblastoma multiforme.

ELIGIBILITY:
- Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Adults over 19 years old
2. Patients with non-small cell lung cancer, metastatic colorectal cancer, metastatic breast cancer, advanced or metastatic kidney cancer, cervical cancer, epithelial ovarian cancer, fallopian tube cancer, primary peritoneal cancer or glioblastoma multiforme.
3. Patients eligible for Zirabev dosage based on local product document, local treatment guidelines and clinical judgment of the medical team.
4. Evidence of a signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

   * Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

1. Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information.
2. Patients for whom Zirabev is contraindicated according to the local product document.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See below
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2025-08-16 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
Safety profile | baseline up to approximately 4 years
  The following items that occurred from the baseline:
  1. Adverse Events (AEs)
  2. Serious Adverse Events (SAEs)
  3. Expected Adverse Events (Expected AEs)
  4. Unexpected Adverse Events (Unexpected AEs)
  5. Adverse Drug Reactions (ADRs)
  6. Serious Adverse Drug Reactions (SADRs)
  7. Expected Adverse Drug Reactions (Expected ADR)
  8. Unexpected Adverse Drug Reactions (Unexpected ADR)

SECONDARY OUTCOMES:
Efficacy profile | baseline up to approximately 4 years
  OR CR SD PD
  1. Non-small cell lung cancer, metastatic colorectal cancer, metastatic breast cancer, advanced or metastatic kidney cancer, cervical cancer, epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
     • Four objective response categories: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) (RECIST 1.1)
  2. Glioblastoma multiforme patients • Four objective response categories: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) (RANO-HGG)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.